CLINICAL TRIAL: NCT06962176
Title: Posterior Mitral Isthmus Line With Vein of Marshall Ethanolisation Compared With Anterior Mitral Lines in Patients With Persistent Atrial Fibrillation
Acronym: MIVANT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Coordinating investigator, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIVANT
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Catheter ablation; Vein of Marshall ethanolization; Mitral line ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Mitral Line Ablation (Experimental): First pulmonary vein isolation (PVI) is performed - either as a first-time isolation (index procedure) or a re-isolation (in repeat procedures). Then a linear lesion is created on the anterior wall of the left atrium, from the roof line to the mitral annulus.
  Interventions: Procedure: Anterior Mitral Line Ablation
- Posterior Mitral Isthmus Ablation with Vein of Marshall Ethanol Infusion (Experimental): As with the anterior approach, pulmonary vein isolation (PVI) is systematically carried out before any additional ablation lines are created - either as initial isolation or re-isolation. In this group the posterior mitral isthmus, a region between the left inferior pulmonary vein and the mitral annulus, is targeted. Endocardial ablation using a dual energy catheter (RF and PF) is combined with ethanol infusion in the vein of Marshall (VOM), which ablates the adjacent epicardial tissue to enhance lesion durability.
  Interventions: Procedure: Posterior Mitral Isthmus Ablation with Vein of Marshall Ethanol Infusion

INTERVENTIONS:
Procedure: Anterior Mitral Line Ablation — First pulmonary vein isolation (PVI) is performed - either as a first-time isolation (index procedure) or a re-isolation (in repeat procedures). Then a linear lesion is created on the anterior wall of the left atrium, from the roof line to the mitral annulus.
  Arms: Anterior Mitral Line Ablation
Procedure: Posterior Mitral Isthmus Ablation with Vein of Marshall Ethanol Infusion — Pulmonary vein isolation (PVI) is systematically carried out before any additional ablation lines are created - either as initial isolation or re-isolation. In this group the posterior mitral isthmus, a region between the left inferior pulmonary vein and the mitral annulus, is targeted. Endocardial ablation using a dual energy catheter (RF and PF) is combined with ethanol infusion in the vein of Marshall (VOM), which ablates the adjacent epicardial tissue to enhance lesion durability.
  Arms: Posterior Mitral Isthmus Ablation with Vein of Marshall Ethanol Infusion

SUMMARY:
The goal of this clinical study is to find out which treatment works best for people with persistent atrial fibrillation (a type of irregular heartbeat). Researchers are comparing two types of heart ablation procedures:

* An anterior mitral line ablation (a treatment at the front part of the heart)
* A posterior mitral line ablation (at the back of the heart), sometimes with an extra step using a small vein called the Vein of Marshall

The main questions the study aims to answer are:

* Which approach works better at fixing the heart rhythm?
* Which approach is safer (less complications)?

People who take part in this study will:

* Undergo an ablation procedure as part of their standard care
* Attend follow-up visits at 1, 3, and 6 months
* Have tests like ECGs, heart ultrasound (echocardiogram), blood tests, heart rhythm monitors (Holter), and a heart CT scan

DETAILED DESCRIPTION:
The MIVANT trial aims to compare two different strategies for treating patients with persistent atrial fibrillation (AF) using catheter ablation techniques. AF is a common heart rhythm disorder, and in persistent forms, it often does not respond adequately to pulmonary vein isolation (PVI) alone. For this reason, many patients require additional ablation lines in the left atrium to reduce arrhythmia recurrence and improve long-term rhythm control.

One such ablation strategy involves creating a linear lesion across the mitral isthmus-a region between the mitral valve and the pulmonary veins. There are two main anatomical approaches to target this area:

* The anterior mitral line, which connects the right superior pulmonary vein to the mitral annulus
* The posterior mitral line, which connects the left inferior pulmonary vein to the mitral annulus

The posterior line is technically more challenging because of the complex anatomy, proximity to blood vessels, and epicardial electrical pathways that can bypass endocardial lesions. However, this difficulty can be addressed by a technique known as Vein of Marshall (VOM) ethanol infusion. The VOM is a small vein near the mitral isthmus that contains nerve fibers and muscle bundles involved in atrial arrhythmias. Infusing ethanol into this vein can help create more effective and lasting ablation lines by reaching areas that standard catheter ablation cannot.

The MIVANT study will enroll 146 adult patients with persistent atrial fibrillation who are already scheduled to receive additional ablation beyond PVI. Patients will be randomized in a 1:1 ratio to undergo either:

* A posterior mitral line ablation, with or without ethanol infusion into the Vein of Marshall, depending on anatomical feasibility
* An anterior mitral line ablation without ethanol infusion

All procedures will be performed under general anesthesia or conscious sedation, using state-of-the-art mapping and ablation tools. Standardized ablation parameters will be followed to ensure consistency and quality across sites.

The main objective of this study is to determine whether the posterior approach-with possible VOM infusion-leads to a higher success rate of procedural bidirectional block across the mitral line, compared to the anterior approach.

Secondary objectives include assessing:

* Safety outcomes such as bleeding, stroke, or coronary artery injury
* Efficiency of the procedure, including total time, fluoroscopy exposure, and number of lesions needed
* Recurrence of atrial arrhythmias at 6 months
* Patient quality of life
* Hospitalizations related to cardiovascular events

Participants will attend follow-up visits at 1, 3, and 6 months, during which they will undergo tests such as ECGs, echocardiography, Holter monitoring, CT coronary angiography, and blood tests.

This study is expected to last a total of 24 months, with 18 months allocated for patient recruitment and a minimum of 6 months follow-up per participant. The study is coordinated by AZ Sint-Jan Brugge AV in Belgium, with possible collaboration from other high-volume centers in France and Switzerland.

The findings of the MIVANT study will help clarify whether posterior mitral isthmus ablation-with the aid of Vein of Marshall ethanolisation-is a more effective and equally safe alternative to the anterior approach in the treatment of persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 years, diagnosed with symptomatic persistent AF with clinical indication for left atrial ablation with a mitral isthmus line. Pulmonary vein will be isolated in all patients before starting the mitral isthmus line (during a previous or the same procedure)

Exclusion Criteria:

* Previous mitral line or any other left atrial ablation beyond pulmonary vein isolation
* Left atrial (LA) thrombus. LA thrombus can be determined by preprocedural imaging: CT, transesophageal echocardiography or MRI.
* LA diameter greater than 60 mm on long axis parasternal view, or left atrial volume more than 250 cc.
* Left ventricular ejection fraction <25%.
* Cardiac surgery within the previous 90 days.
* Expecting cardiac transplantation or other cardiac surgery within 180 days.
* Percutaneous transluminal coronary angioplasty/stenting or myocardial infarction within the previous 30 days.
* Documented history of a thromboembolic event within the previous 60 days.
* Diagnosed atrial myxoma.
* Significant restrictive, constrictive, or chronic obstructive pulmonary disease with chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment
* Women who are pregnant or who plan to become pregnant during the study.
* Acute illness or active infection at time of index procedure
* Renal insufficiency
* Unstable angina.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation.
* Life expectancy less than 1 year.
* Uncontrolled heart failure.
* Presence of a condition that precludes vascular access.
* International normalised ratio (INR) greater than 4 within 24 hours of procedure - for patients taking warfarin.
* Unwilling or unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with procedural linear bidirectional block | During procedure
  After first-pass ablation, bidirectional block across the mitral isthmus line will be assessed by conventional methods consisting of differential pacing maneuvers and documenting widely separated double potentials across the entire length of the line and high-density activation mapping with the Optrell catheter. In the case of absence of block, PF applications will be carried out on the RF line where the earliest activation will be evidenced, for an target index of >550. In the case of absence of block after PF ablation, additional RF and PF ablation points will be performed at the earliest activation sites, adjacent to the previous lesions. A maximum total duration of RF and PF application of 20 min will be allowed for both lines, after which the failure of block will be accepted. Bidirectional conduction block will be reassessed ≥10min after the last ablation lesion along the lines.

SECONDARY OUTCOMES:
Procedural safety | 6 months
  Characterization of complications, including pericardial effusion, stroke and coronary stenosis
Procedural parameters: total procedure time (min) | During procedure
  Comparison of procedural parameters between groups: total procedure time (min)
Procedural parameters: fluoroscopy time (min) | During procedure
  Comparison of procedural parameters between groups: fluoroscopy time (min)
Procedural parameters: total RF ablation time (min) | During procedure
  Comparison of procedural parameters between groups: total RF ablation time
Procedural parameters: total ablation time (min) | During procedure
  Comparison of procedural parameters between groups: total ablation time
Procedural parameters: number of ablation lesions required | During procedure
  Comparison of procedural parameters between groups: number of ablation lesions required
Cardiovascular-related hospitalizations | 6 months
  Characterization of cardiovascular-related hospitalizations in both groups
Recurrence of arrhythmia | 6 months
  Recurrence of arrhythmia, assessed 24 hour Holter monitoring 3 months post procedure and 7-day Holter monitoring 6 months post procedure
Quality of life (SF-36 and AF Symtoms Checklist) | 6 months
  Characterization of quality of life, assessed using the 36-Item Short Form Survey Instrument (SF-36) and the AF Symptom Checklist
Left atrial function at 6 months follow-up | 6 months
  Left atrial function at 6 months follow-up, assessed using transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Jan Brugge AV

IPD SHARING:
Plan to Share IPD: No